CLINICAL TRIAL: NCT05204017
Title: Comprehensive Analysis Platform To Understand, Remedy and Eliminate ALS
Acronym: CAPTURE ALS
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: McGill University (Other); Laval University (Other); University of Toronto (Other); Simon Fraser University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110972
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Progressive Muscular Atrophy; Frontotemporal Degeneration
Keywords: Biomarker; Biorepository; ALS; Disease Progression; MRI; Biofluids
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Muscular Atrophy, Spinal; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA, RNA, Cerebrospinal Fluid, Induced Pluripotent Stem Cells, Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CAPTURE ALS is a long-term data and biorepository platform that will facilitate future ALS research. CAPTURE ALS will provide the standardized systems and tools necessary to collect, store, and analyze vast amounts of multimodal information about ALS. These multimodal datasets and biosamples will be made available for use by researchers or industry across Canada and around the world in accordance with the CAPTURE ALS Data Sharing Policy to advance research on ALS.

DETAILED DESCRIPTION:
In this observational study, participants with ALS and related disorders will be followed longitudinally over the course of a year to examine disease progression. Participants with ALS or a related disorder will have up to 5 in-person visits at screening, 0, 4, 8 and 12 months. Healthy controls are included as comparisons and will have 3 in-person visits at screening, 0 and 8 months. At each visit after screening, patients and healthy controls will undergo an MRI, neurocognitive and speech testing, clinical evaluations specific to ALS (ALSFRS-R, FVC, neurological exam, which are not completed by controls), answer questionnaires about their health and have biospecimens, including blood, saliva and optionally cerebrospinal fluid, collected.

ELIGIBILITY:
[PATIENTS]

Inclusion Criteria:

1. Has ALS, classified as definite, probable, laboratory-supported probable, or possible ALS according to the revised El Escorial criteria or a related neurodegenerative disorder including ALS-FTD, PLS, PMA or asymptomatic individuals with a known ALS mutation (as previously confirmed during regular clinical care)
2. Be of the age of majority in their province of residence/treatment
3. Have the cognitive capacity to provide informed consent
4. Have proficiency in English or French in order to understand study instructions and respond to questionnaires

Exclusion Criteria:

N/A

[HEALTHY CONTROLS]

Inclusion Criteria:

1. Be between the ages of 40-80 unless age matched to a patient (+/-3 years) who is already enrolled
2. Be the age of majority in their province of residence/treatment
3. Have the cognitive capacity to provide informed consent
4. Have proficiency in English of French to understand study instructions and respond to questionnaires

Exclusion Criteria:

1. A history of a neurological disease, including Central Nervous System disease (e.g., stroke, head injury, epilepsy) or Peripheral Nervous System disease (neuropathy, myopathy)
2. A history of psychiatric disease (e.g. depression, bipolar disease) that is clinically diagnosed and/or with the current use of psychiatric medications (e.g. antidepressants) for an indication of a psychiatric disease.
3. Subjects ineligible for an MRI due to a pacemaker or other contraindication according to local MRI policies of the study centre.
4. Significant claustrophobia that would prohibit an MRI (subjects will be required to lie in an MRI scanner for approximately one hour).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with ALS and related motor neuron diseases including ALS-Frontotemporal Dementia (ALS-FTD), Primary Lateral Sclerosis (PLS), Progressive Muscular Atrophy (PMA) and asymptomatic individuals with a known ALS mutation
  AND
  Healthy controls that are age and sex matched to patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) | Once every 4 months for a year
  The ALSFRS-R will be used as a global measure of disease status. It measures activities of daily living and consists of 12 questions, each scored from 0-4, with higher scores representing better function. Changes in ALSFRS-R score over time will be measured.
Forced Vital Capacity (FVC) | Once every 4 months for a year
  FVC will be used as an index of respiratory function over time. FVC is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration.
Speech Testing | Once every 4 months for a year
  Changes in speech function over time will be measured using a web-browser based audio and video data collection tool.
Neurological dysfunction as detected during standard neurological examination | Once every 4 months for a year
  Changes in neurological function over time will be measured through a standard neurological examination.
Magnetic Resonance Imaging (MRI) | Once every 4 months for a year
  Various advanced MRI techniques will be used to assess nervous system structure and function.
Edinburgh Cognitive and Behavioural Screen (ECAS) | Once every 4 months for a year
  Changes in cognitive function over time will be measured by the ECAS.
ALS Assessment Questionnaire (ALSAQ-5) | Once every 4 months for a year
  Changes in quality of life over time will be measured using the ALSAQ-5, a participant reported outcome measure.
World Health Organization Quality of Life Questionnaire (WHO-QOL-BREF) | Once every 4 months for a year
  Changes in quality of life over time will be measured using the WHO-QOL-BREF, a participant reported outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kalra, MD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - University of Toronto / Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University / Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHU de Quebec -Universite de Laval, Québec, Quebec

REFERENCES:
- [Derived] Saunders N, Magnussen C, Kang H, Blais M, Bhinder H, Pfeffer G, Genuis SK, Bouvier L, Anand T, Abou-Haidar R, Abrahao A, Boivin MN, Bowser R, Bubela T, Chiappini J, Das S, Dhanoa A, Dupre N, Evans A, Ferry N, Frater Y, Genge A, Graham SJ, Greiner R, Medina YI, Johnston WS, Jones KE, Karamchandani J, Kriz J, Luth W, Matte G, Rogaeva E, Robertson J, Seres P, Tam F, Taylor D, Tremblay-Desbiens C, Velde CV, Yunusova Y, Zinman L, Kalra S. Comprehensive analysis platform to understand, remedy, and eliminate amyotrophic lateral sclerosis (CAPTURE ALS): Study protocol for a Canadian multicenter, multimodal, longitudinal observational study. PLoS One. 2025 Dec 4;20(12):e0332430. doi: 10.1371/journal.pone.0332430. eCollection 2025. PMID 41343582